CLINICAL TRIAL: NCT07208266
Title: Contingency Management as a Behavioral Intervention for Patients With Opioid Use Disorder : Implementation and Efficacy in the Inpatient Setting at Assiut University Hospital.
Brief Title: Contingency Management for Opioid Use Disorder in Inpatients at Assiut University Hospital
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ragaei Raouf Zaki Samuel, Resident doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuroPsych-CM-2025
Record Dates: First submitted 2025-09-18; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder (OUD)
Keywords: Opioid Use Disorder; Contingency Management; Assiut University Hospital
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency Management Intervention (Experimental)
  Interventions: Behavioral: contingency management

INTERVENTIONS:
Behavioral: contingency management — Participants with opioid use disorder admitted to the inpatient addiction management unit will receive a contingency management (CM) program as a behavioral intervention. The program consists of providing positive reinforcement (small rewards or incentives) contingent upon objective evidence of desired behaviors, primarily drug abstinence verified by urine toxicology screening. The intervention will be delivered throughout the inpatient stay (approximately two weeks). Participants' adherence and abstinence will be monitored, and rewards will be adjusted based on performance.

SUMMARY:
A scientific study to design and implement a contingency management (CM) program, and to evaluate its effectiveness in promoting abstinence and treatment adherence among individuals with opioid use disorder, as well as to explore its potential for broader implementation in clinical settings.

DETAILED DESCRIPTION:
Addiction and drug use can have negative consequences on the health, economy, productivity, and social aspects of communities. Addictive disorders are of high prevalence and often associated with other psychiatric and somatic diseases. Severe cases, often complicated by multiple dependencies of substances and advanced stages of the disease can require the involvement of a variety of caregivers, who are requested to sufficiently cooperate and interact to guarantee an optimal outcome of treatment. Tolerance and withdrawal are the two hallmark criteria of physiological addiction, and, arguably, may also be considered as aspects of a more general concept of preoccupation (or as features that contribute to preoccupation). Tolerance refers to the need to engage in the behavior at a relatively greater level than in the past to achieve previous levels of appetitive effects. As tolerance increases, one likely spends more time locating and engaging in an addiction. Thus, tolerance may indicate increasing preoccupation. Withdrawal refers to physiological or acquired discomfort experienced upon abrupt termination of an addictive behavior. If withdrawal symptoms exist, and worsen, one is likely to be spending more and more time recovering from the after-effects of the addiction, and focused in thought and action on how to cope (e.g., by using again). That is, one is more preoccupied with the addiction when one is spending more time locating, engaging, and recovering from that behavior, and this may reflect processes of tolerance and withdrawal. Historically, addiction treatment systems and research have been organized to provide and improve the outcomes of acute episodes of care. The conceptual model has been that an addicted person seeks treatment, completes an assessment, receives treatment, and is discharged, all in a period of weeks or months. This orientation stands at variance with clinical experience and studies conducted over several decades, which confirm that, although some individuals can be successfully treated within an acute care framework, more than half the patients entering publicly funded addiction programs require multiple episodes of treatment over several years to achieve and sustain recovery. The progress of many patients is marked by cycles of recovery, relapse, and repeated treatments, often spanning many years before eventuating in stable recovery, permanent disability, or death.

Contingency management (CM) is a promising intervention for treating drug dependence. CM treatments rearrange the environment to detect drug use readily and to promote participation in activities that are inconsistent with drug use. These treatments encourage participation upon objective evidence of drug abstinence or engagement in non-drug-related activities. Contingency management (CM) is a behavioral intervention where reinforcement is provided when biologically confirmed drug abstinence is demonstrated, typically in the form of a urine test. Unlike some substance use disorders (SUDs) where there are pharmacological treatments available, all empirically supported treatments for stimulant use disorder are behavioral, and contingency management (CM) has the strongest support. CM, or the provision of reinforcement to encourage abstinence from substances or other behaviors, has strong empirical support, established over decades of research, for the treatment of SUDs, including stimulant, nicotine, alcohol, and opioid use disorders. Although CM is efficacious, it is rarely implemented in practice. A primary obstacle is cost.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Have a diagnosis of a substance use disorder (SUD) according to DSM-5 criteria
* Be able to understand and provide informed consent
* Be willing to comply with study procedures, including regular drug screening and attendance tracking
* Must be able to swallow tablets

Exclusion Criteria:

* Have a severe cognitive impairment or active psychosis that interferes with participation
* Currently experiencing a medical condition that would make participation unsafe

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 55 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Relapse Risk Assessment: Assessed using the Advance Warning of Relapse (AWARE) Questionnaire administered at program entry and exit. Changes in AWARE scores will indicate changes in relapse risk and warning signs. | From baseline (admission) until discharge (~2 weeks), and at 3 months post-discharge
Proportion of opioid-negative urine drug screens during inpatient stay and at 3-month follow-up | From baseline (admission) until discharge (~2 weeks), and at 3 months post-discharge

REFERENCES:
- [Background] Rawson RA, Erath TG, Chalk M, Clark HW, McDaid C, Wattenberg SA, Roll JM, McDonell MG, Parent S, Freese TE. Contingency Management for Stimulant Use Disorder: Progress, Challenges, and Recommendations. J Ambul Care Manage. 2023 Apr-Jun 01;46(2):152-159. doi: 10.1097/JAC.0000000000000450. Epub 2023 Feb 3. PMID 36745163
- [Background] Kwon M, Yang S, Park K, Kim DJ. Factors that affect substance users' suicidal behavior: a view from the Addiction Severity Index in Korea. Ann Gen Psychiatry. 2013 Nov 12;12(1):35. doi: 10.1186/1744-859X-12-35. PMID 24220264
- [Background] Petry NM, Barry D, Alessi SM, Rounsaville BJ, Carroll KM. A randomized trial adapting contingency management targets based on initial abstinence status of cocaine-dependent patients. J Consult Clin Psychol. 2012 Apr;80(2):276-85. doi: 10.1037/a0026883. Epub 2012 Jan 9. PMID 22229758
- [Background] Coughlin LN, Zhang L, Frost MC, Khazanov G, McKay JR, DePhilippis D, Lin LA. Contingency management for substance use disorders in the U.S. Veterans Health Administration: 2018-2022. J Subst Use Addict Treat. 2024 Aug;163:209400. doi: 10.1016/j.josat.2024.209400. Epub 2024 May 11. PMID 38735480
- [Background] McDonell MG, Skalisky J, Burduli E, Foote A Sr, Granbois A, Smoker K, Hirchak K, Herron J, Ries RK, Echo-Hawk A, Barbosa-Leiker C, Buchwald D, Roll J, McPherson SM. The rewarding recovery study: a randomized controlled trial of incentives for alcohol and drug abstinence with a rural American Indian community. Addiction. 2021 Jun;116(6):1569-1579. doi: 10.1111/add.15349. Epub 2021 Jan 14. PMID 33220122
- [Background] Petry NM, Tedford J, Austin M, Nich C, Carroll KM, Rounsaville BJ. Prize reinforcement contingency management for treating cocaine users: how low can we go, and with whom? Addiction. 2004 Mar;99(3):349-60. doi: 10.1111/j.1360-0443.2003.00642.x. PMID 14982548
- [Background] Dennis M, Scott CK. Managing addiction as a chronic condition. Addict Sci Clin Pract. 2007 Dec;4(1):45-55. doi: 10.1151/ascp074145. PMID 18292710
- [Background] Sussman S, Sussman AN. Considering the definition of addiction. Int J Environ Res Public Health. 2011 Oct;8(10):4025-38. doi: 10.3390/ijerph8104025. Epub 2011 Oct 20. PMID 22073026
- [Background] Hofer D, Wenger F, Kohler M, Badertscher M. [Addiction in psychiatric ambulatory service]. Ther Umsch. 2014 Oct;71(10):609-16. doi: 10.1024/0040-5930/a000600. German. PMID 25257115
- [Background] GBD 2016 Alcohol and Drug Use Collaborators. The global burden of disease attributable to alcohol and drug use in 195 countries and territories, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Psychiatry. 2018 Dec;5(12):987-1012. doi: 10.1016/S2215-0366(18)30337-7. Epub 2018 Nov 1. PMID 30392731
- See also: Related Info — https://bmcpsychology.biomedcentral.com/articles/10.1186/s40359-025-02638-8#citeas
- See also: Related Info — https://case.edu/socialwork/centerforebp/sites/default/files/2024-11/CM%20for%20OUD%20Research%20Summary%20Report%2011.22.24.pdf